CLINICAL TRIAL: NCT05408624
Title: Pilot Study Evaluating Outpatient Management of Tubo-ovarian Abscesses
Acronym: AmbATO
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC21_0011
Record Dates: First submitted 2022-05-23; First posted 2022-06-07 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Abscess; Pelvic Inflammatory Disease; Pelvic Infection
Keywords: Tubo-ovarian abscess; pelvic inflammatory disease; antibiotics; outpatient management; ultrasound-guided transvaginal drainage; laparoscopy
MeSH Terms: conditions — Abscess; Pelvic Inflammatory Disease; Pelvic Infection | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- prospective group - ultrasound transvaginal drainage: Patients with TOA with ultrasound-guided transvaginal drainage with outpatient management
  Interventions: Procedure: ultrasound transvaginal drainage
- retrospective group - ultrasound transvaginal drainage: Patients with TOA in 2016, 2017 and 2018 with ultrasound-guided transvaginal drainage in conventional hospitalization
  Interventions: Procedure: ultrasound transvaginal drainage
- retrospective group - laparoscopy: Patients with TOA in 2016, 2017 and 2018 with laparoscopy in conventional hospitalization
  Interventions: Procedure: laparoscopy

INTERVENTIONS:
Procedure: ultrasound transvaginal drainage — Ultrasound-guided transvaginal drainage of TOA by a puncture under simple sedation or analgesia with/or under general anesthesia
  Groups: prospective group - ultrasound transvaginal drainage; retrospective group - ultrasound transvaginal drainage
Procedure: laparoscopy — Laparoscopy for drainage of TOA under general anesthesia
  Groups: retrospective group - laparoscopy

SUMMARY:
Pelvic inflammatory diseases (PID) require antibiotic treatment. Among PID, the investigators distinguish: pelvi-peritonitis and pelvic collections such as Douglas abscess and/or tubo-ovarian abscess (TOA).

Recent recommendations published in December 2018 by the National College of French Gynecologists and Obstetricians (CNGOF) suggest that it is preferable to drain TOA when their size is greater than 3-4 cm. Ultrasound-guided transvaginal drainage is recommended as first-line treatment because of its ease of performance and its effectiveness. In the literature, many authors have demonstrated the feasibility and efficacy of transvaginal drainage associated with antibiotics in the treatment of TOA. Since ultrasound-guided transvaginal drainage is a less invasive alternative therapeutic procedure than laparoscopy for the drainage of TOA, it would be compatible with outpatient management. This mode of management can be carried out in a dedicated outpatient or functional exploration room with the help of a nurse but without an anesthetic team present. This gesture is simple and short-lived. In addition, the antibiotics used have pharmacological properties allowing oral intake from their initiation.

The investigators have proposed a new service protocol to treat TOA in this outpatient mode. The investigators therefore wish to analyze this new protocol from these three angles: 1/ the feasibility of this care, 2/ the quality of life of the patients through questionnaires given throughout the care and 3/ an evaluation of the 'efficiency.

DETAILED DESCRIPTION:
Pelvic inflammatory diseases (PID) require antibiotic treatment. Among PID, the investigators distinguish: pelvi-peritonitis and pelvic collections such as Douglas abscess and/or tubo-ovarian abscess (TOA).

Recent recommendations published in December 2018 by the National College of French Gynecologists and Obstetricians (CNGOF) suggest that it is preferable to drain TOA when their size is greater than 3-4 cm. Ultrasound-guided transvaginal drainage is recommended as first-line treatment because of its ease of performance and its effectiveness. In the literature, many authors have demonstrated the feasibility and efficacy of transvaginal drainage associated with antibiotics in the treatment of TOA. Since ultrasound-guided transvaginal drainage is a less invasive alternative therapeutic procedure than laparoscopy for the drainage of TOA, it would be compatible with outpatient management. This mode of management can be carried out in a dedicated outpatient or functional exploration room with the help of a nurse but without an anesthetic team present. This gesture is simple and short-lived. In addition, the antibiotics used have pharmacological properties allowing oral intake from their initiation.

The investigators have proposed a new service protocol to treat TOA in this outpatient mode. The investigators therefore wish to analyze this new protocol from these three angles: 1/ the feasibility of this care, 2/ the quality of life of the patients through questionnaires given throughout the care and 3/ an evaluation of the 'efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Major patient at the time of inclusion
* Patient with diagnosis of TOA with a latero-uterine mass measuring at least 3 cm

Exclusion Criteria:

* Patient with severity criteria requiring hospitalization:

  * Clinical severity criteria: haemodynamically unstable patient, septic shock, defense or contracture, sepsis, pelviperitonitis
  * Comorbidities: diabetic imbalance, curative anticoagulation
* Patient with a formal indication for laparoscopy:

  * Diagnostic doubt with suspicion of an associated oncological or digestive pathology
  * Presence of an intra-abdominal intrauterine device (IUD)
  * Abscess not accessible vaginally
* Patient who does not meet the eligibility criteria for outpatient hospitalization defined by French High Autority of Health
* Patient under guardianship or curatorship
* Patient does not speak French
* Patient not benefiting from social security coverage
* Current pregnancy
* Confirmed allergy to one of the antibiotics (ceftriaxone, metronidazole or doxycycline)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with diagnosis of TOA with a latero-uterine mass measuring at least 3 cm
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Cure rate | one month
  The cure rate is defined by a composite criterion at 1 month of the procedure:
  * Apyrexia (temperature <38,0°c)
  * Absence of re-intervention for pelvic collection (TOA) in the month following the transvaginal drainage
  * Absence of second-line antibiotic therapy, extension, new antibiotic in the month following the transvaginal drainage

SECONDARY OUTCOMES:
eligibility | 2 years
  Number of patients included in the protocol compared to the number of eligible patients
Discharge | 2 years
  Discharge from hospital within 24 hours of the drainage
Rehospitalization | 1 month
  Rehospitalization: reason, duration and care
Measure of Pain | 1 month
  Pain is assessed by Numerical Rating Scale (NRS) (0-10). Absence of pain (EN=0/10), mild pain (EN<4/10), absence of metrorrhagia and absence of leucorrhoea
residual mass | 1 month
  Absence of residual mass ≥ 3cm on pelvic ultrasound
complications | 1 month
  Presence of complications (digestive, urinary, parietal)
antibiotic therapy | 1 month
  Change of antibiotic therapy (except adequate adaptation to the antibiogram). Change of antibiotic therapy is assessed by the need to add another antibiotic with a broader spectrum of action, following a poor clinical or biological evolution.
Quality of life with EQ-5D-5L | 1 month
  Satisfaction and Quality of life completed by the patients on the day of the drainage before the procedure, at 48 hours and at 1 month
Quality of life with Medical Outcome Study Short Form 12 (SF12) | 1 month
  Satisfaction and Quality of life, questionnaires completed by the patients on the day of the drainage before the procedure, at 48 hours and at 1 month.
  Each question is assessed on a Likert scale, with 5 to 6 possible levels of response possible responses. The 8 dimensions combine synthetic information to calculate a physical composite score (PCS) and a mental score (SCP) and a mental composite score (SCM). The higher the score, the greater the patient's ability.
Quality of life with Patient Global Impression of Improvement (PGI-I) questionnaires | 1 month
  Satisfaction and Quality of life , questionnaires completed by the patients on the day of the drainage before the procedure, at 48 hours and at 1 month The PGI-I is a transition scale that is a single question asking the patient to rate their urinary tract condition now, as compared with how it was prior to before beginning treatment on a scale from 1. Very much better to 7. Very much worse.
Evaluation of the direct costs | 1 month
  Evaluation of the direct costs of care for the 3 treatment strategies for complicated IGH of the ATO type, according to a time horizon of 1 month and a collective perspective

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nantes, Nantes, France